CLINICAL TRIAL: NCT06443658
Title: Benefits of Inhalation of Hypertonic Saline Solution Prior to ELTGOL Physiotherapy in Bronchiectasis
Brief Title: Benefits of Inhalation of Hypertonic Saline Solution Prior to Physiotherapy ELTGOL Technique in Bronchiectasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Collaborators: University Hospital of Girona Dr. Josep Trueta (Network); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FISHT2021
Record Dates: First submitted 2024-01-23; First posted 2024-06-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Bronchiectasis Adult
Keywords: airway clearance; hypertonic saline; respiratory physiotherapy
MeSH Terms: interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ELTGOL group (Other): Control group. Patients will do twice-daily ELTGOL technique
  Interventions: Other: ELTGOL
- ELTGOL + isotonic saline solution (0,9%) (Placebo Comparator): Placebo group. Patients will do twice-daily ELTGOL technique and will receive 5ml of 0.9% saline before performing the ELTGOL technique in the morning
  Interventions: Drug: Isotonic saline; Other: ELTGOL
- ELTGOL + hypertonic saline solution (7%) (Experimental): Experimental group. Patients will do twice-daily ELTGOL technique and will receive 5ml of 7% saline before performing the ELTGOL technique in the morning
  Interventions: Other: Hypertonic saline; Other: ELTGOL

INTERVENTIONS:
Other: Hypertonic saline — Patients from intervention group will inhale hypertonic saline solution 5 minutes before performing the morning ELTGOL technique
  Arms: ELTGOL + hypertonic saline solution (7%)
Drug: Isotonic saline — Patients from placebo group will inhale isotonic saline solution 5 minutes before performing the morning ELTGOL technique
  Other Names: Physiologic saline
  Arms: ELTGOL + isotonic saline solution (0,9%)
Other: ELTGOL — Patients from control group will perform the ELTGOL technique twice-daily

SUMMARY:
Bronchiectasis is a chronic bronchial disease in which the usual capacity to remove secretions does not function correctly, causing mucus retention that leads to chronic infection. As with all infections, the use of antibiotics and puss removal are essential treatment elements. Physiotherapeutic techniques are used to assist in the removal of secretions, although these are time-consuming practices that need to be much better studied and which patients often do not continue practicing diligently. A physiotherapeutic technique called (Slow prolonged expiration in lateral decubitus) ELTGOL has been shown to be somewhat effective but as the mucus is viscous in this disorder, it can be difficult to get it to move. It is thought that saline solution inhalations may reduce mucus viscosity and could help to ease expectoration, facilitating the removal of the mucus by the physiotherapeutic technique. This project aims to test this hypothesis, which if true could represent an advance in the treatment of this severely debilitating disease.

DETAILED DESCRIPTION:
Bronchiectasis is a prevalent chronic infectious disease with impaired mucociliary clearance. The persistence of high bacterial loads in the bronchi is associated with airway and systemic inflammation. Management is based on treatment of bronchial infection and on removal of secretions by airway clearance techniques (ACTs) although no therapy has been approved due to low quality of evidence. Inhalation of hypertonic saline (HS) could be useful in facilitate mucus removal especially if it is administer prior an effective ACT.Our hypothesis is that the long-term combination of HS and the ELTGOL technique will facilitate secretion removal in bronchiectasis and this will be associated with changes in mucus composition and better control of the disease.

Study design: A 12-month parallel-group, multicentre, double-blind randomised-controlled trial. Patients will be randomly assigned to receiving HS, isotonic saline (IS) or no inhalation before practicing ELTGOL technique.

The main objective is to evaluate the effect of the combination of once-daily inhaled HS and twice daily ELTGOL technique in mucus clearance in bronchiectasis. Secondary aims: to determine its effect on mucus properties, the impact of cough,exacerbations, quality of life, microbiology and pulmonary function; to evaluate adverse effects and adherence.

Study population: adult patients with non-cystic fibrosis bronchiectasis in stable state with chronic mucopurulent or purulent sputum.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with bronchiectasis confirmed by high resolution computed tomography
* No exacerbations in the previous month
* Chronic mucopurulent and purulent sputum
* ≥10ml daily expectoration
* At least one exacerbation in the previous year
* (Forced expiratory volume the 1st second) FEV1 ≥30% after bronchodilation
* Sign the informed consent

Exclusion Criteria:

* Current smokers or a smoking history of ≥20 p-y
* Asthma, allergic bronchopulmonary aspergillosis or Cystic Fibrosis
* Pregnant or lactating women
* Following mucoactive treatment in the previous month
* Inability to perform ELTGOL, spirometry or to attend visits
* Practicing pulmonary rehabilitation in the previous 6 months
* Change of treatment the previous month
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The change in the sputum weight in grams during intervention | Baseline and 12 months later
  Sputum weight will be measured with a precision balance after the intervention

SECONDARY OUTCOMES:
Change in sputum properties 1 | Changes between Month 1 and Month 12
  Sputum properties will be evaluated analyzing viscosity (mPa/s) and elasticity (Pa)
Change in sputum properties 2 | Changes between Month 1 and Month 12
  Sputum properties will be evaluated analyzing solids in sputum
Change from baseline in the 24hours sputum volume in milliliters | Over the 12-month treatment period.
  Sputum volume will be measured with a calibrated container
Change from baseline in the 24hours sputum weight | Over the 12-month treatment period.
  Sputum weight will be measured with a precision balance
Change in cough | Over the 12-month treatment period.
  Assessed with the Leicester Cough Questionnaire (LCQ). Score form 3 to 21 (3 better and 21 worse cough)
Number of exacerbations | Over the 12-month treatment period.
  Based on clinical history
Time to the first exacerbation | Over the 12-month treatment period.
  Based on clinical history
Change in quality of life | Over the 12-month treatment period
  Assessed with Bronchiectasis health questionnaire (BHQ). BHQ score from 0-100 (0 best and 100 worse quality of life)
Change in post-bronchodilator ( forced expiratory volume at one second) FEV1 | Over the 12-month treatment period in ml
  Assessed with a forced spirometry
Treatment adherence 1 | Over the 12-month treatment period
  Assessed through vial counting.
Treatment adherence 2 | Over the 12-month treatment period
  Assessed through the diary card.
Treatment adherence 3 | Over the 12-month treatment period
  Assessed through Morisky-Green test. Score from 0 to 4 (0 best and 4 worse adherence)
Adverse events 1 | Over the 12-month treatment period
  Assessed by Borg scale at the end of interventions. Score 0-10 (0 best and 10 worse breathlessness)
Adverse events 2 | Over the 12-month treatment period
  Assessed by oxygen desaturation
Adverse events 3 | Over the 12-month treatment period
  Assessed by Visual Analogue Scale (VAS) scale (pain assessment)
Change in sputum weight during intervention | Between Month 12 and Month 13
  Sputum weight will be measured with a precision balance after the intervention
Change in sputum volume in 24h sputum volume | Between Month 12 and Month 13
  Sputum volume will be measured with a calibrated container
Change in cough | Between Month 12 and Month 13
  Assessed with the Leicester Cough Questionnaire (LCQ). Score form 3 to 21 (3 better and 21 worse cough)
Change in post-bronchodilator FEV1 | Between Month 12 and Month 13
  Assessed with a forced spirometry
Change in quality of life | Between Month 12 and Month 13
  Assessed with Bronchiectasis health questionnaire (BHQ). BHQ score from 0-100 (0 best and 100 worse quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Vendrell, PhD MD, Principal Investigator — University Hospital of Girona Dr. Josep Trueta
Locations (1):
- University Hospital of Girona Dr. Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected data can be shared as long as it is for research collaboration
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the manuscript is accepted for publication
Access Criteria: Study data access will be provided for collaborative purposes

REFERENCES:
- [Background] Munoz G, de Gracia J, Buxo M, Alvarez A, Vendrell M. Long-term benefits of airway clearance in bronchiectasis: a randomised placebo-controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701926. doi: 10.1183/13993003.01926-2017. Print 2018 Jan. PMID 29326318
- [Background] Munoz G, Buxo M, de Gracia J, Olveira C, Martinez-Garcia MA, Giron R, Polverino E, Alvarez A, Birring SS, Vendrell M. Validation of a Spanish version of the Leicester Cough Questionnaire in non-cystic fibrosis bronchiectasis. Chron Respir Dis. 2016 May;13(2):128-36. doi: 10.1177/1479972316632005. Epub 2016 Feb 22. PMID 26902541